CLINICAL TRIAL: NCT06495086
Title: A High-Flow Nasal Cannula Versus Noninvasive Ventilation in Acute Exacerbations of Chronic Obstructive Pulmonary Disease: A Single-blind Randomized Trial
Brief Title: HFNC vs. NIV in Acute COPD Exacerbations
Acronym: HFNCstdy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 137-2023
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: COPD Exacerbations; Acute Hypercapnic Respiratory Failure; Respiratory Failure
Keywords: High-flow nasal cannula; Noninvasive ventilation; COPD exacerbations; efficacy; safety
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Single center
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this single-blind study, we assigned the participants randomly to one of three treatment groups using a computer-generated randomization program (SAS Institute, 1990). Each participant was assigned an identification number indicating their treatment group. An experienced clinician, who was blinded to the null hypothesis and did not participate in the evaluation of results, administered the treatments and recorded patient data on a pre-prepared case data form.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- NIV group (Active Comparator): The NIV group received bilevel-positive airway pressure.
  Interventions: Device: NIV
- HFNC-30 group (Active Comparator): HFNC-30 group received HFNC therapy at flow rates of 30 L/min.
  Interventions: Device: HFNC-30
- HFNC-50 group (Active Comparator): HFNC-50 group received HFNC therapy at flow rates of 50 L/min.
  Interventions: Device: HFNC-50

INTERVENTIONS:
Device: NIV — The NIV group received bilevel-positive airway pressure. During NIV, the tidal volume was set to 6-8 mL/kg, positive expiratory end pressure (PEEP) to 3-5 cm H2O, and pressure support ventilation (PSV) to 8-12 cm H2O by a clinician with 8 years of experience. To reduce potential bias, the clinician was blinded to the null hypothesis.
  Arms: NIV group
Device: HFNC-30 — The HFNC-30 group received HFNC therapy at flow rates of 30 L/min. During HFNC, the humidifier was set to an open position, the heated air temperature was maintained at 37°C, and the FiO2 was adjusted to maintain an oxygen saturation (SpO2) measured via pulse oximetry of at least 92%.
  Arms: HFNC-30 group
Device: HFNC-50 — The HFNC-50 group received HFNC therapy at flow rates of 50 L/min. During HFNC, the humidifier was set to an open position, the heated air temperature was maintained at 37°C, and the FiO2 was adjusted to maintain an oxygen saturation (SpO2) measured via pulse oximetry of at least 92%.
  Arms: HFNC-50 group

SUMMARY:
The investigators investigated the efficacy and safety of High Flow Nasal Cannula (HFNC) at different flow rates compared to non-invasive ventilation (NIV) in patients presenting to the emergency department (ED) with acute exacerbations of Chronic obstructive pulmonary disease (COPD) who did not respond adequately to bronchodilator therapy and continued to exhibit hypercapnic respiratory failure. Specifically, the investigators tested the hypothesis that HFNC would be more effective at reducing partial pressure of carbon dioxide (PaCO2) levels and hospital stay duration and would be associated with greater patient comfort than NIV.

DETAILED DESCRIPTION:
The patients were divided randomly into one of three study groups: NIV, HFNC-30, and HFNC-50. The investigators collected patient data, including demographic characteristics (age and sex), vital signs upon admission (systolic blood pressure [SBP], respiratory rate [RR], and heart rate [HR]), complaints and symptoms upon admission, initial arterial blood gas parameters (e.g., pH, PaCO2, lactate, and bicarbonate), length of stay, ED revisits, patient satisfaction, intubation status, and clinical outcomes (hospitalization, admission to the intensive care unit [ICU], or 28-day mortality). Changes in arterial blood gas parameters (e.g., ΔpH, ΔPaCO2, Δlactate, and Δbicarbonate) before treatment vs. 30, 60, and 120 minutes after treatment were recorded using a pre-prepared case data form.

ELIGIBILITY:
Inclusion Criteria:

- patients age ≥18 years with a confirmed diagnosis of COPD who presented to the ED with exacerbations that did not respond to bronchodilator therapy

Exclusion Criteria:

* patients aged younger than 18 years
* patients had an arterial pH ≤ 7.25;
* patients were in cardiopulmonary arrest;
* patients had unstable cardiac arrhythmias or hemodynamic instability;
* patients showed persistent hypoxemia despite supplemental oxygen therapy;
* patients were unconscious or uncooperative;
* patients could not protect their airway or manage secretions;
* patients had cardiogenic pulmonary edema, active hemoptysis, pneumothorax, recent upper respiratory tract/esophagus surgery, significant airway obstruction (e.g., laryngeal mass or tracheal tumor), active upper gastrointestinal bleeding, or facial trauma or deformities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in pH in arterial blood gas before vs. after treatment | at 30, 60, and 120 minutes relative to baseline
  The investigators assessed the changes in pH before treatments vs. 30, 60, and 120 minutes after treatments.
Changes in PaCO2 in arterial blood gas before vs. after treatment | at 30, 60, and 120 minutes relative to baseline
  The investigators assessed the changes in PaCO2 before treatments vs. 30, 60, and 120 minutes after treatments.
Changes in lactate in arterial blood gas before vs. after treatment | at 30, 60, and 120 minutes relative to baseline
  The investigators assessed the changes in lactate before treatments vs. 30, 60, and 120 minutes after treatments.
Changes in bicarbonate in arterial blood gas before vs. after treatment | at 30, 60, and 120 minutes relative to baseline
  The investigators assessed the changes in bicarbonate before treatments vs. 30, 60, and 120 minutes after treatments.

SECONDARY OUTCOMES:
Assessing the need for rescue treatment and treatment-related complications | 120 minutes after initial treatment
  The investigators assessed the need for invasive respiratory support and also evaluated treatment-related complications.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, M.D., Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Rezaei A, Fakharian A, Ghorbani F, Idani E, Abedini A, Jamaati H. Comparison of high-flow oxygenation with noninvasive ventilation in COPD exacerbation: A crossover clinical trial. Clin Respir J. 2021 Apr;15(4):420-429. doi: 10.1111/crj.13315. Epub 2020 Dec 22. PMID 33269553
- [Result] Liu S, Walline JH, Zhu H, Li Y, Wang C, Liu J. High-flow nasal cannula therapy with sequential noninvasive ventilation versus noninvasive ventilation alone as the initial ventilatory strategy in acute COPD exacerbations: study protocol for a randomized controlled trial. Trials. 2022 Dec 29;23(1):1060. doi: 10.1186/s13063-022-06963-w. PMID 36581995
- [Result] Cortegiani A, Longhini F, Madotto F, Groff P, Scala R, Crimi C, Carlucci A, Bruni A, Garofalo E, Raineri SM, Tonelli R, Comellini V, Lupia E, Vetrugno L, Clini E, Giarratano A, Nava S, Navalesi P, Gregoretti C; H. F.-AECOPD study investigators. High flow nasal therapy versus noninvasive ventilation as initial ventilatory strategy in COPD exacerbation: a multicenter non-inferiority randomized trial. Crit Care. 2020 Dec 14;24(1):692. doi: 10.1186/s13054-020-03409-0. PMID 33317579
- [Result] Rittayamai N, Phuangchoei P, Tscheikuna J, Praphruetkit N, Brochard L. Effects of high-flow nasal cannula and non-invasive ventilation on inspiratory effort in hypercapnic patients with chronic obstructive pulmonary disease: a preliminary study. Ann Intensive Care. 2019 Oct 22;9(1):122. doi: 10.1186/s13613-019-0597-5. PMID 31641959
- [Derived] Haciosman O, Ergenc H, Az A, Dogan Y, Sogut O. A high-flow nasal cannula versus noninvasive ventilation in acute exacerbations of chronic obstructive pulmonary disease. Am J Emerg Med. 2025 Jan;87:38-43. doi: 10.1016/j.ajem.2024.10.043. Epub 2024 Oct 28. PMID 39481328